CLINICAL TRIAL: NCT00700986
Title: A Randomised, Double-Blind, Placebo-Controlled, 2-Period Cross-Over Study in Healthy Male Volunteers, to Investigate Retinal Function Following a Single 800mg Oral Dose of AZD9056
Brief Title: Cross-over Study to Investigate Retinal Function Following Administration of a Single Dose of AZD9056
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Dr Mark Layton MD, MRCP (UK), Medicine Science Director, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: D1520C00020; EUDRACT No. 2008-000752-27
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Electroretinography; Rheumatoid Arthritis; Anti-TNF; Disease Modifying Anti-Rheumatic Drugs (DMARD)
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — AZD9056

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD9056
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD9056 — Oral tablet, 800mg, one single administration
  Arms: 1
Drug: Placebo — Single dose
  Arms: 2

SUMMARY:
The purpose of the study is to determine whether treatment with a single 800mg dose of AZD9056, a medication which has been developed as a possible treatment for Rheumatoid Arthritis, has an effect on the function of the retina

ELIGIBILITY:
Inclusion Criteria:

* Volunteers must be able to undergo the Electroretinography assessments
* Volunteers must have an intra ocular pressure of less than 25mmHg and 6/6 vision

Exclusion Criteria:

* Volunteers must pass a test that assesses whether they are at risk of narrow angle glaucoma
* Volunteers must not a family history of colour blindness, they must also pass a colour blindness test
* Volunteers must not have a history or current neurological or opthalmological (eye) disease

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2008-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
The effect of a single dose of AZD9056 (800mg) on retinal function will be assessed by Electroretinography | Electroretinography measurements will be performed at baseline, 6 hours post dosing at both treatment and crossover placebo treatment visits, and at post study medical follow up visits.

SECONDARY OUTCOMES:
The effect of a single dose of AZD9056 (800mg) on retinal function will be assessed by measurements of visual acuity, contrast sensitivity and colour vision. | Visual acuity, contrast sensitivity and colour vision measurements will be performed at a training visit, at baseline, 2.5 hours post dosing at both treatment and crossover placebo treatment visits, and at post study medical follow up visits.
The effect of a single dose of AZD9056 (800mg) on occipital function will be assessed by measurements of visual evoked potential. | Visual evoked potential measurements will be performed at a training visit, at baseline, 4 hours post dosing at both treatment and crossover placebo treatment visits, and at post study medical follow up visits.
The effect of a single dose of AZD9056 (800mg) on cognitive function will be assessed by psychomotor testing. | Psychomotor testing will be performed at a training visit, at baseline, 8.5 and 24 hours post dosing at both treatment and crossover placebo treatment visits, and at post study medical follow up visits.

CONTACTS AND LOCATIONS:
Overall Officials: William Fahy, MA, MBBS (Hons), Principal Investigator — AstraZeneca Clinical Pharmacology Unit, Nottingham; Mark Layton, MD, MRCP (UK), Study Director — AstraZeneca Alderley Park
Locations (1):
- Research Site, Nottingham, Nottinghamshire, United Kingdom